CLINICAL TRIAL: NCT04130464
Title: The Impact of the Continuous Infusion of Intraperitoneal Analgesics on Postoperative Pain After Minimally Invasive Hysterectomy: a Randomized Controlled Trial
Brief Title: Intraperitoneal Infusion of Analgesic for Postoperative Pain Management
Acronym: ON-Q
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ying Liu (Other)
Collaborators: Avanos Medical (Other)
Responsible Party: Sponsor-Investigator, Ying Liu, PI, George Washington University
Organization: George Washington University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 180423
Record Dates: First submitted 2019-10-16; First posted 2019-10-17 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Hysterectomy; Gynecologic Surgical Procedures; Narcotic Use; Pain, Postoperative
Keywords: Intraperitoneal; Pain Pump; Ropivacaine; Ketorolac Tromethamine
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Ketorolac Tromethamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study; the surgeon and the patient will not know which study group they are a part of. Only the IDS pharmacist and IDS pharmacy technician will know which group each study patient has been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ropivacaine (Experimental): Subjects will receive a continuous intraperitoneal infusion of ropivacaine
  Interventions: Drug: Ropivacaine Infusion from ON-Q Pump
- Ropivacaine + Ketorolac (Experimental): Subjects will receive a continuous intraperitoneal infusion of ropivacaine + ketorolac
  Interventions: Drug: Ropivacaine + Ketorolac Infusion from ON-Q Pump
- Normal Saline (Placebo Comparator): Subjects will receive a continuous intraperitoneal infusion of normal saline
  Interventions: Drug: Normal Saline Infusion from ON-Q Pump

INTERVENTIONS:
Drug: Ropivacaine Infusion from ON-Q Pump — Infusion of 0.2% ropivacaine at 8 mL/hour for 72 hours
  Other Names: Naropin
  Arms: Ropivacaine
Drug: Ropivacaine + Ketorolac Infusion from ON-Q Pump — Infusion of 0.2% ropivacaine + 30 mg ketorolac at 8 mL/hour for 72 hours
  Other Names: Naropin; Toradol
  Arms: Ropivacaine + Ketorolac
Drug: Normal Saline Infusion from ON-Q Pump — Infusion of 0.9% normal saline at 8 mL/hour for 72 hours
  Other Names: Saline solution
  Arms: Normal Saline

SUMMARY:
The study is a prospective, double-blinded, placebo-controlled multi-center trial to measure if postoperative pain and the amount of narcotics used are reduced by a clinically significant amount in women undergoing minimally invasive hysterectomy receiving a continuous infusion of intraperitoneal (IP) local anesthetic (LA) or a continuous infusion of LA combined with an NSAID compared with a control group who receives only 0.9% normal saline.

DETAILED DESCRIPTION:
* Any patient desiring minimally invasive hysterectomy will be contacted by a study team member during their visit to the MIGS (minimally invasive gynecologic surgery) clinic. The risks and benefits of participation will be explained to them. If they choose to participate they will sign the consent form at that time or if they need more time to consider participation they will sign later. They will then complete the health-related quality of life (HrQoL) questionnaire UFS-QOL* before surgery.
* Computer-generated randomization will be used to randomize patients between 3 groups:
* Group A: receiving a continuous infusion of intraperitoneal local anesthetic (LA) during 72 hours
* Group B: receiving a continuous infusion of intraperitoneal LA combined with an NSAID during 72 hours
* Group C: receiving a continuous infusion of intraperitoneal placebo during 72 hours.
* Study participants will then undergo a minimally invasive hysterectomy by one of the highly experienced minimally invasive gynecologists using a standard technique. At the conclusion of the procedure, all women will have an infusion catheter attached to an ON-Q pump inserted percutaneously into the pelvis under direct laparoscopic vision. The catheter tip will be placed in the peritoneal cavity at the vaginal vault. In order to ensure patency of the catheter tubing, a 10 mL bolus of assigned medication will be given. The ON-Q pump infusion will then provide 540 mL of assigned medication for a total of 72 hours following surgery.
* Surgical variables (length of surgery, estimated blood loss, type of analgesia and anesthesia used, concomitant procedures, uterine weight, ASA, and intraoperative complications - organ injury (bladder, bowel, vaginal laceration), EBL > 1000 cc, conversion to laparotomy, transfusion) will be recorded on a data collection sheet.
* Additional analgesia will be administered by the nursing staff in the PACU at the patient's request. The total dose of analgesia over the 72 postoperative hours will be calculated for each woman (e.g. each of the following was considered to be one dose; 1 g of paracetamol, 50 mg diclofenac, 400 mg ibuprofen, 50 mg tramadol). The total morphine equivalents per patient will also be recorded.
* All medication administered for pain as well as VAS pain scores at 1, 2, 4, 6, 24, 48, and 72 hours postoperatively will be recorded.
* Subjects will be discharged when clinically appropriate and according to our usual hospital procedure, which is usually same day discharge. Subjects staying in hospital for less than 72 hours will be given verbal and written instructions on catheter removal.
* The subjects will be given a post-operative pain diary to fill out during their 2 week recovery period including pain scores and amount of pain medication used. This diary will be collected at their first post-operative visit at around 2 weeks postoperatively. Subjects will be asked to complete the EQ-5D again during this visit. Postoperative complications will also be recorded (ICU-admission, reoperation, transfusion, DVT/PE, readmission, bowel obstruction/ileus, incision seroma/cellulitis/hematoma/separation/hernia, and cuff cellulitis/abscess/dehiscence/granulation tissue).
* Hospital (operative and pathology reports) and clinical (clinical visit notes) reports will be reviewed to compare baseline demographics, past surgical history, past medical history, comorbidities, and complications between groups.
* Pumps and syringes will be filled with study drugs depending on the assigned group to a max of 540 mL for pumps and a max of 10 mL for syringes:
* Group A: receiving a continuous infusion of intraperitoneal local anesthetic (LA) during 72 hours: 10 mL bolus of 0.2% Ropivacaine + 540 mL of 0.2% Ropivacaine at 8 mL/hour infusion
* Group B: receiving a continuous infusion of intraperitoneal LA combined with an NSAID during 72 hours: 10 mL bolus of 0.2% Ropivacaine combined with 30mg/550mL toradol + 540 mL of 0.2% Ropivacaine combined with 30mg/550mL toradol at 8 mL/hour infusion
* Group C: receiving a continuous infusion of intraperitoneal placebo during 72 hours: 10 mL bolus of 0.9% normal saline + 540 mL of 0.9% normal saline at 8 mL/hour infusion
* The IDS research pharmacist will fill the pumps for use and a member of the research team will transport the filled pumps to the hospital for the surgeries.
* Statistical Analysis: Pre-operative variables such as patient demographic and clinical information (medical and surgical history) will be recorded and compared as well as intra-operative variables such as surgical modality, length of surgery, estimated blood loss, concomitant procedures, uterine weight, ASA, and complications. Before and after their surgery, patients will complete a questionnaire regarding quality of life and pain. To combine the results of both sites, REDCap will be used to securely share de-identified data. These outcome variables will be analyzed by calculating the unadjusted and adjusted means and 95% confidence intervals using simple and multiple linear regressions.

ELIGIBILITY:
Inclusion Criteria:

* Hysterectomy planned for a benign gynecologic reason (no evidence of, or concern for, malignancy in the cervix, uterus, tubes or ovaries. Benign gynecologic reasons to have a hysterectomy include fibroids, abnormal uterine bleeding, endometriosis, and pelvic pain.)
* Patient is scheduled to have surgery with a fellowship trained minimally invasive gynecologic surgeons at one of the study sites.
* Patient is planned for a robotic assisted total laparoscopic hysterectomy (RA-TLH) or a total laparoscopic hysterectomy (TLH).
* Patient is capable of informed consent.
* Patient is capable of completing the questionnaires.

Exclusion Criteria:

* Concern for malignancy
* The procedure is scheduled outside MIGS department.
* Allergy to any study related medication (i.e. Ketorolac and Ropivacaine)
* Patient is enrolled in another pain management study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Pain Level 1 Hour Postoperative | 1 hour postoperative
  Rating from 0 "No pain sensation" to 10 "most intense pain imaginable"
Pain Level 2 Hours Postoperative | 2 hours postoperative
  Rating from 0 "No pain sensation" to 10 "most intense pain imaginable"
Pain Level 4 Hours Postoperative | 4 hours postoperative
  Rating from 0 "No pain sensation" to 10 "most intense pain imaginable"
Pain Level 6 Hours Postoperative | 6 hours postoperative
  Rating from 0 "No pain sensation" to 10 "most intense pain imaginable"
Pain Level 24 Hours Postoperative | 24 hours postoperative
  Rating from 0 "No pain sensation" to 10 "most intense pain imaginable"
Pain Level 48 Hours Postoperative | 48 hours postoperative
  Rating from 0 "No pain sensation" to 10 "most intense pain imaginable"
Pain Level 72 Hours Postoperative | 72 hours postoperative
  Rating from 0 "No pain sensation" to 10 "most intense pain imaginable"

SECONDARY OUTCOMES:
The total dose of analgesics taken over the 72 postoperative hours | Within 72 hours postoperative
  Each of the following was considered to be one dose: 1 g of paracetamol, 50 mg diclofenac, 400 mg ibuprofen, 50 mg tramadol

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Keller, MD, Principal Investigator — Physician
Locations (2):
- United States (2):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - The GW Medical Faculty Associates, Washington D.C., District of Columbia